CLINICAL TRIAL: NCT05669573
Title: Safety of 6 Hours Feeding After Extracorporeal Shock Wave Lithotripsy of Pancreatic Stone: a Multicentre, Open-label, Randomized, Controlled Trial
Brief Title: Safety of 6 Hours Feeding After Extracorporeal Shock Wave Lithotripsy of Pancreatic Stone
Acronym: SHEEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Pudong New Area Gongli Hospital (Other); First People's Hospital of Hangzhou (Other); LanZhou University (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHEEL202210
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Duct Stone; ESWL; Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding group (Experimental): Patients in the early diet group started oral intake 6 hours after ESWL of the day of procedure with a soft diet comprised 200 mL with 170 kilocalories. Observe closely until 24h, and then continue to fasting until the next ESWL/ERCP or change the diet to the general diet according to the actual clinical needs.
  Interventions: Procedure: Early feeding group
- Standard fasting group (Active Comparator): Patients in the standard fasting group were fasted for 24 hours after the first ESWL operation, and close observation during this fasting period. After 24 hours, according to the actual clinical needs, continue to fast until the next ESWL/ERCP operation, or change the diet to a general diet.
  Interventions: Procedure: Standard fasting group

INTERVENTIONS:
Procedure: Early feeding group — Patients in the early diet group started oral intake 6 hours after ESWL of the day of procedure with a soft diet comprised 200 mL with 170 kilocalories.
  Arms: Early feeding group
Procedure: Standard fasting group — Patients in the standard fasting group were fasted for 24 hours after the first ESWL operation, and close observation during this fasting period.
  Arms: Standard fasting group

SUMMARY:
The purpose of this study is to evaluate the safety of eating 6 hours after Extracorporeal Shock Wave Lithotripsy (ESWL). At present, ESWL and Endoscopic Retrograde Cholangiopancreatography (ERCP) are the routine ways to treat pancreatic duct stones. For large stones (diameter > 5mm) , ESWL often needs to be performed many times. In clinical practice, fasting for 24 hours after surgery is often used, but long-term fasting brings strong discomfort to patients. However, the consensus for initiation timing of oral nutrition has not yet been established after ESWL. Thus, we design this trial to evaluate the safety of early feeding based on 6 hours parameter instead of the consensus definition.

DETAILED DESCRIPTION:
In recent years, studies have shown that early recovery of enteral nutrition has significant benefits for patients. Early recovery of oral feeding and drinking as well as early oral supplementary nutrition after surgery can promote the recovery of intestinal motor function, help maintain intestinal mucosal function, prevent postoperative flora disorder and diarrhea, shorten postoperative hospital stay, and improve postoperative anxiety of patients.This study mainly evaluated the safety of feeding 6 hours after ESWL, including the risk of post-ESWL pancreatitis and other adverse events, as well as the length of hospital stay, medical expenses, pain, etc. This research conclusion is helpful to provide more scientific and reasonable fasting time for patients after ESWL, improve patient comfort, reduce the risk of adverse events, shorten hospital stay, save medical expenses, and guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis who completed ESWL.

Exclusion Criteria:

* Readmitted to the hospital during enrollment of the study;
* Cannot eat or rely on jejunal nutrition tube to give total parenteral nutrition for various reasons;
* With acute pancreatitis, perforation, infection, bleeding, steinstrasse and other complications and other serious clinical adverse events within 6 hours after ESWL;
* Suspected or confirmed malignancy
* Pancreatic ascites;
* Coagulation dysfunction;
* Taking chemotherapy drugs and immunosuppressants for a long time;
* Acute pancreatitis exacerbation or acute exacerbation of chronic pancreatitis (including biliary pancreatitis);
* Pregnant or breastfeeding women;
* Patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
the incidence of post-ESWL pancreatitis | within 24 hours after ESWL
  A diagnosis of post-ESWL pancreatitis was thus made if two of three of the following criteria were met, in accordance with the revised Atlanta international consensus: pain consistent with pancreatitis; amylase or lipase of at least three times the upper normal limit within 24 h of the procedure; or characteristic findings on imaging.

SECONDARY OUTCOMES:
the severity of post-ESWL pancreatitis | within 24 hours after ESWL
  stratified as mild, moderate, or severe, mainly on the basis of length of hospitalisation and need for invasive treatment
the incidence of other post-ESWL complications | within 24 hours after ESWL
  Other post ESWL complications includes bleeding, infection, steinstrasse, and perforation.
the transient adverse events | within 24 hours after ESWL
  Transient adverse events were defined as transient injuries caused by shock waves that required no medical intervention and did not prolong hospitalisation, including asymptomatic hyperamylasaemia, haematuria, and acute gastrointestinal mucosal injury (eg, haematemesis, melena, or haematochezia) caused by ESWL.
abdominal pain relief rate | within 24 hours after ESWL
  Use the Visual Analogue Scale (VAS). VAS can be calculated ranging from 0 (no pain) to 10 (severe pain).
hunger relief rate | within 24 hours after ESWL
  Use the Visual Analogue Scale (VAS). VAS can be calculated ranging from 0 (not hungry at all) to 10 (hungriest possible).

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao L, Liu Y, Xie T, Wang T, Guo HL, Pan J, Wang D, Bi YW, Ji JT, Xin L, Du TT, Lin JH, Zhang D, Zeng XP, Zou WB, Chen H, Li BR, Liao Z, Cong ZJ, Shi RH, Li ZS, Hu LH. Risk Factors and Nomogram for Pancreatic Stone Formation in Chronic Pancreatitis over a Long-Term Course: A Cohort of 2,153 Patients. Digestion. 2020;101(4):473-483. doi: 10.1159/000500941. Epub 2019 Jun 25. PMID 31238312